CLINICAL TRIAL: NCT02401958
Title: Acute Effect of Resistance Training in Inflammatory Markers in Women With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Carolina Pereira Nunes Pinto, Physiotherapist, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP UNIFESP -
Record Dates: First submitted 2015-03-19; First posted 2015-03-30 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rheumatoid Arthritis Group (Experimental): Resistance Training
  Interventions: Other: Resistance training
- Healthy control Group (Active Comparator): Resistance Training
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — 17 volunteers with RA and 17 without the disease, with a mean age of 54.7 + 6.63 underwent a resistance exercise session with a set of 12 repetitions at 50% of one repetition maximum (1RM ) and a set of 8 repetitions at 75% of 1RM. The exercises performed were: knee extension, knee flexion, hip abduction and hip adduction. Blood samples were obtained 30 minutes before, 5 minutes before, immediately after, 1 hour, 2 hours and 24 hours after the exercise session.

SUMMARY:
ABSTRACT Introduction: Rheumatoid arthritis (RA) is a systemic inflammatory, chronic and progressive disease that can lead to joint destruction and important functional disability. Chronic inflammation, with a substantial increase in the amount of pro-inflammatory cytokines in synovial joint, is one of the biggest challenges in controlling RA. Resistance exercise has been recognized for positively modulate inflammation in healthy subjects. Objective: To evaluate the effect of an acute bout of resistance exercise on serum concentrations of tumor necrosis factor alpha (TNF-α), interleukin 1 receptor antagonist(IL-1ra), interleukin 1 beta (IL-1β), C reactive protein (CRP), interleukin 6 (IL-6), interleukin 10 (IL-10), and cartilage oligomeric matrix protein (COMP) in postmenopausal women with RA and women without the disease. Methods: 17 volunteers with RA and 17 without the disease, with a mean age of 54.7 + 6.63 underwent a resistance exercise session with a set of 12 repetitions at 50% of one repetition maximum (1RM ) and a set of 8 repetitions at 75% of 1RM. The exercises performed were: knee extension, knee flexion, hip abduction and hip adduction. Blood samples were obtained 30 minutes before, 5 minutes before, immediately after, 1 hour, 2 hours and 24 hours after the exercise session. Serum glucose concentrations prior to exercise were also measured. The investigators used the Student's't test, the model of analysis of variance with repeated measures and Bonferroni method of multiple comparisons to analyze the data, being considered statistically significant levels of p <0.05.

ELIGIBILITY:
*Rheumatoid Arthritis Group

Inclusion Criteria:

* Women classified acording to the American College of Rheumatology's criteria to rheumatoid arthritis
* Post menopausal women
* Stable medication three months before study

Exclusion Criteria:

* Women with rheumatoid arthritis with functional class IV, acording to ACR criteria
* Women engaged in some type of regular exercise program;
* Failure: heart, coronary, respiratory, renal and / or hepatic (uncompensated);
* Uncompensated systemic hypertension;
* Volunteers with other associated inflammatory diseases;
* Unable to perform the exercises.

  * Control group We included in the control group of this study postmenopausal volunteers, without Rheumatoid Arthritis. Exclusion criteria were the same as those adopted for the participants of the Rheumatoid Arthritis Group

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in one (or more) of the inflammatory markers | 30 minutes before training; 5 minutes before training; 5 minutes after training; 1 hour after training; 2 hours after training; 24 hours after training
  TNF-alfa, IL1-beta, IL1-ra, PCR, IL10, IL6

SECONDARY OUTCOMES:
No change in inflammatory markers | 30 minutes before training; 5 minutes before training; 5 minutes after training; 1 hour after training; 2 hours after training; 24 hours after training
  TNF-alfa, IL1-beta, IL1-ra, PCR, IL10, IL6

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil